CLINICAL TRIAL: NCT06719245
Title: Prevention of PostAmputation Pain With Targeted Muscle Reinnervation: A National, Multicenter, Randomized, Sham-controlled Superiority Trial, Comparing Standard Neurectomy With Targeted Muscle Reinnervation in Amputations of the Lower Extremities
Brief Title: Prevention of PostAmputation Pain With Targeted Muscle Reinnervation
Acronym: PreventPAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Alrijne Hospital (Other); Medical Center Haaglanden (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); UMC Utrecht (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other); Isala (Other)
Responsible Party: Principal Investigator, jlgroen, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL87196.058.24
Record Dates: First submitted 2024-07-12; First posted 2024-12-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Amputation, Surgical; Phantom Limb Pain; Neuroma Amputation; Surgery
Keywords: TMR; Amputation; Phantom pain; Neuroma
MeSH Terms: conditions — Phantom Limb; Neuroma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Neurectomy (control) (Other): Standard Neurectomy during amputation (control)
  Interventions: Procedure: Standard neurectomy
- Targeted Muscle Reinnervation (intervention) (Other): Targeted Muscle Reinnervation (TMR) during amputation (intervention)
  Interventions: Procedure: Targeted Muscle Reinnervation (TMR)

INTERVENTIONS:
Procedure: Targeted Muscle Reinnervation (TMR) — In short: each transected nerve is identified after amputation and is dissected proximally for length. A nerve stimulator is used to identify functional motor nerve branches. Near the point where the motor branch enters the muscle, the motor nerve branch is transected and an end-to-end coaptation is performed with a nearby amputated nerve.
  Arms: Targeted Muscle Reinnervation (intervention)
Procedure: Standard neurectomy — During the amputation a standard neurectomy will be performed based on the surgeons preference. Standard neurectomy will include cutting of the nerve, with or without traction, with or without coagulation, and with or without infiltration with a local anesthetic (i.e., ropivacaine) or phenol. Ligation of the nerve will not be allowed.
  Arms: Standard Neurectomy (control)

SUMMARY:
The goal of this study is to compare postamputation pain (phantom limb pain and residual limb pain) one year postoperatively in patients who received a lower extremity amputation (LEA) with standard nerve handling (neurectomy) versus those who received Targeted Muscle Reinnervation (TMR).

Patients between 18 and 75 years old, scheduled for an LEA (transfemoral to transtibial) as a primary or secondary sequela of vascular disease, are randomized into standard neurectomy or TMR. TMR is a frequently studied surgical technique and prevents neuroma formation by rerouting a cut mixed nerve end to a functional motor nerve.

The investigators hypothesize that TMR during amputation surgery will significant improve PostAmputation Pain (PAP), quality of life, participation in family life and society, and reduction of health-related costs. Participants will be asked to complete multiple online questionnaires postoperatively regarding these outcomes at five evaluation moments (at 2 weeks, and at 3, 6, 9, and 12 months).

DETAILED DESCRIPTION:
Rationale: In the Netherlands, approximately 3300 lower extremity amputations (sacroiliac to forefoot) are performed each year. In current amputation practice, the nerves are simply cut, without employing any nerve surgical techniques to prevent the development of chronic pain due to neuroma formation. Around 61% of these patients develop postamputation pain (PAP). PAP is a severe lifelong disabling condition profoundly affecting quality of life.

Microsurgical nerve handling can prevent the formation of a painful neuroma and its sequelae. In recent years, targeted muscle reinnervation (TMR) has been the most frequently studied technique with promising results. TMR prevents neuroma formation by rerouting a cut mixed nerve end to a functional motor nerve.

The expected benefit of the implementation of TMR during amputation surgery is a significant reduction in the incidence of PAP. Prevention of this chronic pain syndrome will lead to a significant improvement in quality of life, participation in family life and society, and reduction of health-related costs for thousands of amputation patients every year. To achieve this, a transformation of nerve handling during amputation is needed.

Objective: To compare postamputation pain (phantom limb pain and residual limb pain) one year postoperatively in patients who received a lower extremity amputation (LEA) with standard nerve handling (neurectomy) versus those who received TMR.

Study design: A national, multicenter, randomized, sham-controlled superiority trial, comparing standard neurectomy with TMR in amputations of the lower extremities.

Study population: Patients between 18 and 75 years old, scheduled for an LEA (transfemoral to transtibial) as a primary or secondary sequela of vascular disease.

Intervention: Patients with an LEA are randomized into standard neurectomy or TMR. TMR in short: each transected nerve is identified after amputation and is dissected proximally for length. A nerve stimulator is used to identify functional motor nerve branches. Near the point where the motor branch enters the muscle, the motor nerve branch is transected, and an end-to-end coaptation is performed with a nearby amputated nerve.

Main study parameters: The mean difference in pain scores for phantom limb pain and residual limb pain one year postoperatively. Pain is measured for 30 consecutive days (Pain Diary) on the 11-point (0-10) numerical rating scale (NRS) and according to the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Behavior and Interference Questionnaire Short Forms (7a and 8a, respectively).

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: The additional risks of performing TMR during amputation are negligible. TMR can be performed at any level of the lower extremities with a standardized technique. For TMR to be possible, in upper leg amputations, an additional incision (ca 10 centimetres) has to be made on the dorsal side of the leg, medial tot the sartorius muscle. In our experience this will not result in more postoperative pain or difficulty in sitting. To properly blind study participants this additional incision for upper leg amputations must also be superficially performed in the control group. Another factor that will differ from current standards is that the procedure will take 30 to 90 minutes longer. The extra time investment will depend on technical aspects related to the level of amputation and surgeon experience. Although an increase in surgical time of this length is associated with a slightly higher risk of infection, studies have not found more complications in patients undergoing acute TMR compared to those receiving standard care. The burden of the study is minimal, as participation only requires patients to fill out multiple online questionnaires at five evaluation moments (at 2 weeks, and at 3, 6, 9, and 12 months). Prophylactic TMR results in a reduction of the chance to develop PAP. The risks and the burden for patients are negligible.

ELIGIBILITY:
Inclusion criteria

* Patients aged between 18 and 75 years old.
* Scheduled for a transtibial, through-knee, or transfemoral amputation as a primary or secondary sequela of vascular disease.

Exclusion criteria

* Insensate limbs at the level of amputation.
* Complex Regional Pain Syndrome.
* Existing neuroma or prior neuroma surgery in the affected limb.
* Undergoing radiotherapy on the affected limb.
* Cognitive impairment, or delirium at the time of consent.
* Patients who are unfit for general anesthesia.
* No nerve surgeon trained in the TMR procedure is available

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative residual limb pain | at 12 months
  Postoperative residual limb pain will be scored on the 11-point (0-10) Numeric Rating Scale (NRS) for 30 consecutive days in a pain diary. A higher score indicates more pain.
Postoperative phantom limb pain | at 12 months
  Postoperative phantom limb pain will be scored on the 11-point (0-10) Numeric Rating Scale (NRS) for 30 consecutive days in a pain diary. A higher score indicates more pain.
Postoperative pain behavior | at 12 months
  Postoperative pain behavior will be scored using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Behavior Short Form 7a. The results will be scored on a scale from 7 to 35 points, with a higher score indicating that pain has a greater influence on behavior.
Postoperative pain interference | at 12 months
  Postoperative pain interference will be scored using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form 8a. The results will be scored on a scale from 8 to 40 points, where a higher score indicates greater interference of pain with daily life

SECONDARY OUTCOMES:
Postoperative residual limb pain | at 3, 6, and 9 months
  Postoperative residual limb pain will be scored on the 11-point (0-10) Numeric Rating Scale (NRS) at one timepoint. A higher score indicates more pain.
Postoperative phantom limb pain | at 3, 6, and 9 months
  Postoperative phantom limb pain will be scored on the 11-point (0-10) Numeric Rating Scale (NRS) at one timepoint. A higher score indicates more pain.
Postoperative pain behavior | at 3, 6, and 9 months
  Postoperative pain behavior will be scored using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Behavior Short Form 7a. The results will be scored on a scale from 7 to 35 points, with a higher score indicating that pain has a greater influence on behavior.
Postoperative pain interference | at 3, 6, and 9 months
  Postoperative pain interference will be scored using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form 8a. The results will be scored on a scale from 8 to 40 points, where a higher score indicates greater interference of pain with daily life
Neuropathic pain | at 12 months
  Using the Neuropathic pain component in chronic pain syndromes (PainDetect) questionnaire. The results will be scored on a scale from 0 to 38. A higher score indicates a greater likelihood of experiencing neuropathic pain
Hospital anxiety | at 12 months
  Using the Hospital Anxiety and Depression Scale (HADS). The results will be scored on a scale from 0 to 21. A higher score indicates a greater likelihood of experiencing anxiety
Depression | at 12 months
  Using the Hospital Anxiety and Depression Scale (HADS). The results will be scored on a scale from 0 to 21. A higher score indicates a greater likelihood of experiencing depression.
Global perceived effect | at 12 months
  Using the Global Perceived effect (GPE-DV) questionnaire to evaluate the patients' view on recovery and satisfaction of the treatment.
Prosthetic rehabilitation | at 12 months
  Measured with the Prosthetic Limb Users Survey of Mobility (PLUS-M, seven items short form). The results will be scored on a scale from 7 to 35. A higher score indicates a better prosthetic rehabilitation.
EuroQol-5D-5L | at 2 weeks, and at 3, 6, 9 and 12 months
  Quality of life using the EuroQol-5D-5L questionnaire. A higher score indicates worse quality of life.
Medical consumption costs | at 3, 6, 9, and 12 months
  Cost effectiveness analysis with a trial-based cost-utility analysis from a societal perspective (i.e., cost per QALY). Using the Medical Consumption Questionnaire (iMCQ)
Productivity costs | at 3, 6, 9, and 12 months
  Cost effectiveness analysis with a trial-based cost-utility analysis from a societal perspective (i.e., cost per QALY). Using the Productivity Costs Questionnaire (iPCQ)
Budget impact analysis (BIA). | at 12 months
  Budget impact analysis using the ZonMW BIA tool to estimate the financial impact of different implementation scenarios at the national level
Pain medication use | at 3, 6, 9, and 12 months
  The Medication Quantification Scale measures the extent of pain medication use. A higher score indicates an increased use or dosage of pain medication.
Type of pain | at 3, 6, 9 and 12 months
  Type of pain (local, diffuse, radiating) will be reported using the pain sketches from the Interdisciplinary Care for Amputees Network (ICAN).

OTHER OUTCOMES:
Surgical time | at 0 months
  Surgical time measured in minutes
Length of hospital stay | at 0 months
  Postoperative length of stay in the hospital
Adverse events | 30 days postoperative
  i.e., infection, rebleed. Scored with the Clavien-Dindo score form 1 to 5. A higher score indicates a more severe complication.

CONTACTS AND LOCATIONS:
Overall Officials: Justus L Groen, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (7):
- Netherlands (7):
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - Isala Zwolle, Zwolle, Overijssel
  - Leiden University Medical Center, Leiden, South Holland
  - Alrijne Zorggroep, Leiderdorp, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Haaglanden Medisch Centrum, The Hague, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
By embracing the FAIR principles (Findability, Accessibility, Interoperability and Reusability of digital assets), we underscore our commitment to robust, transparent, and ethically sound scientific practices that advance research integrity and propel scientific progress. Using the Leiden University Medical Center (LUMC) Data Management Tool, with support of the LUMC section of Advanced Data Management we ensure that our data is findable, enabling easy discovery through well-structured metadata and standardized identifiers. Through our commitment to accessibility, we guarantee that both researchers and the broader community can access our data with minimal barriers, fostering collaboration and knowledge dissemination. Interoperability remains a focal point, as we structure our data in standardized formats and utilize established vocabularies, facilitating seamless integration with other datasets and tools. Our dedication to reusability ensures that the data generated through our trial
Supporting Information: Study Protocol
Time Frame: After completion of the study, the key file will be archived in the hospital's study documentation on a protected location on the network hard drive for 15 years in accordance with article 17 of the European good clinical practice directive.
Access Criteria: Before acquiring the deidentified individual patient data used in the results of the published work related to this protocol (incl. tables, figures, supplementary files), researcher must sign a data sharing agreement. Data will made available to those who submit a reasonable request with a methodologically sound proposal.

REFERENCES:
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Mioton LM, Dumanian GA, Shah N, Qiu CS, Ertl WJ, Potter BK, Souza JM, Valerio IL, Ko JH, Jordan SW. Targeted Muscle Reinnervation Improves Residual Limb Pain, Phantom Limb Pain, and Limb Function: A Prospective Study of 33 Major Limb Amputees. Clin Orthop Relat Res. 2020 Sep;478(9):2161-2167. doi: 10.1097/CORR.0000000000001323. PMID 32452928
- [Background] Dal-Re R, Janiaud P, Ioannidis JPA. Real-world evidence: How pragmatic are randomized controlled trials labeled as pragmatic? BMC Med. 2018 Apr 3;16(1):49. doi: 10.1186/s12916-018-1038-2. PMID 29615035
- [Background] Torrance N, Lawson KD, Afolabi E, Bennett MI, Serpell MG, Dunn KM, Smith BH. Estimating the burden of disease in chronic pain with and without neuropathic characteristics: does the choice between the EQ-5D and SF-6D matter? Pain. 2014 Oct;155(10):1996-2004. doi: 10.1016/j.pain.2014.07.001. Epub 2014 Jul 11. PMID 25020004
- [Background] Parsons B, Schaefer C, Mann R, Sadosky A, Daniel S, Nalamachu S, Stacey BR, Nieshoff EC, Tuchman M, Anschel A. Economic and humanistic burden of post-trauma and post-surgical neuropathic pain among adults in the United States. J Pain Res. 2013 Jun 17;6:459-69. doi: 10.2147/JPR.S44939. Print 2013. PMID 23825931
- [Background] Groffen AJ, Klapwijk T, van Rootselaar AF, Groen JL, Tijssen MA. Genetic and phenotypic heterogeneity in sporadic and familial forms of paroxysmal dyskinesia. J Neurol. 2013 Jan;260(1):93-9. doi: 10.1007/s00415-012-6592-5. Epub 2012 Jun 30. PMID 22752065
- [Background] Valerio IL, Dumanian GA, Jordan SW, Mioton LM, Bowen JB, West JM, Porter K, Ko JH, Souza JM, Potter BK. Preemptive Treatment of Phantom and Residual Limb Pain with Targeted Muscle Reinnervation at the Time of Major Limb Amputation. J Am Coll Surg. 2019 Mar;228(3):217-226. doi: 10.1016/j.jamcollsurg.2018.12.015. Epub 2019 Jan 8. PMID 30634038
- [Background] Frantz TL, Everhart JS, West JM, Ly TV, Phieffer LS, Valerio IL. Targeted Muscle Reinnervation at the Time of Major Limb Amputation in Traumatic Amputees: Early Experience of an Effective Treatment Strategy to Improve Pain. JB JS Open Access. 2020 May 6;5(2):e0067. doi: 10.2106/JBJS.OA.19.00067. eCollection 2020 Apr-Jun. PMID 33123667
- [Background] Malessy MJA, de Boer R, Munoz Romero I, Eekhof JLA, van Zwet EW, Kliot M, Dahan A, Pondaag W. Predictive value of a diagnostic block in focal nerve injury with neuropathic pain when surgery is considered. PLoS One. 2018 Sep 12;13(9):e0203345. doi: 10.1371/journal.pone.0203345. eCollection 2018. PMID 30208078
- [Background] Deeyor ST, Kisana HM, Hui CH, Stecher C, Hustedt JW. Targeted Muscle Reinnervation Does Not Increase the Risk of Postsurgical Complication or Overall Cost. Plast Reconstr Surg Glob Open. 2022 Aug 24;10(8):e4488. doi: 10.1097/GOX.0000000000004488. eCollection 2022 Aug. PMID 36032374
- [Background] Schwingler PM, Moman RN, Hunt C, Ashmore Z, Ogletree SP, Uvodich ME, Murad MH, Hooten WM. Prevalence of postamputation pain and its subtypes: a meta-analysis with meta-regression. Pain Rep. 2021 May 4;6(1):e918. doi: 10.1097/PR9.0000000000000918. eCollection 2021. PMID 33981935
- [Background] Poyntz SA, Hacking NM, Dalal M, Fowler S. Peripheral Interventions for Painful Stump Neuromas of the Lower Limb: A Systematic Review. Clin J Pain. 2018 Mar;34(3):285-295. doi: 10.1097/AJP.0000000000000533. PMID 28678059
- [Background] Dumanian GA, Potter BK, Mioton LM, Ko JH, Cheesborough JE, Souza JM, Ertl WJ, Tintle SM, Nanos GP, Valerio IL, Kuiken TA, Apkarian AV, Porter K, Jordan SW. Targeted Muscle Reinnervation Treats Neuroma and Phantom Pain in Major Limb Amputees: A Randomized Clinical Trial. Ann Surg. 2019 Aug;270(2):238-246. doi: 10.1097/SLA.0000000000003088. PMID 30371518
- [Background] Berger LE, Shin S, Haffner ZK, Huffman SS, Spoer DL, Sayyed AA, Franzoni G, Bekeny JC, Attinger CE, Kleiber GM. The application of targeted muscle reinnervation in lower extremity amputations: A systematic review. Microsurgery. 2023 Oct;43(7):736-747. doi: 10.1002/micr.31030. Epub 2023 Mar 2. PMID 36864779
- [Background] Walsh AR, Lu J, Rodriguez E, Diamond S, Sultan SM. The Current State of Targeted Muscle Reinnervation: A Systematic Review. J Reconstr Microsurg. 2023 Mar;39(3):238-244. doi: 10.1055/s-0042-1755262. Epub 2022 Aug 21. PMID 35988579
- [Background] Chang BL, Hill AL, Mondshine J, Harbour PW, Episalla NC, Attinger CE, Kleiber GM. Primary Targeted Muscle Reinnervation in Above-Knee Amputations in Patients with Unsalvageable Limbs from Limb-Threatening Ischemia or Infection. J Reconstr Microsurg. 2024 Feb;40(2):109-117. doi: 10.1055/a-2086-0395. Epub 2023 May 4. PMID 37142250
- [Background] Ives GC, Kung TA, Nghiem BT, Ursu DC, Brown DL, Cederna PS, Kemp SWP. Current State of the Surgical Treatment of Terminal Neuromas. Neurosurgery. 2018 Sep 1;83(3):354-364. doi: 10.1093/neuros/nyx500. PMID 29053875
- [Background] Dellon AL, Mackinnon SE. Treatment of the painful neuroma by neuroma resection and muscle implantation. Plast Reconstr Surg. 1986 Mar;77(3):427-38. doi: 10.1097/00006534-198603000-00016. PMID 2937074
- [Background] Alexander JH, Jordan SW, West JM, Compston A, Fugitt J, Bowen JB, Dumanian GA, Pollock R, Mayerson JL, Scharschmidt TJ, Valerio IL. Targeted muscle reinnervation in oncologic amputees: Early experience of a novel institutional protocol. J Surg Oncol. 2019 Sep;120(3):348-358. doi: 10.1002/jso.25586. Epub 2019 Jun 13. PMID 31197851
- [Background] O'Brien AL, Jordan SW, West JM, Mioton LM, Dumanian GA, Valerio IL. Targeted Muscle Reinnervation at the Time of Upper-Extremity Amputation for the Treatment of Pain Severity and Symptoms. J Hand Surg Am. 2021 Jan;46(1):72.e1-72.e10. doi: 10.1016/j.jhsa.2020.08.014. Epub 2020 Oct 22. PMID 33268236
- [Background] O'Brien AL, West JM, Gokun Y, Janse S, Schulz SA, Valerio IL, Moore AM. Longitudinal Durability of Patient-Reported Pain Outcomes after Targeted Muscle Reinnervation at the Time of Major Limb Amputation. J Am Coll Surg. 2022 May 1;234(5):883-889. doi: 10.1097/XCS.0000000000000117. PMID 35426401
- [Background] Kang NV, Woollard A, Michno DA, Al-Ajam Y, Tan J, Hansen E. A consecutive series of targeted muscle reinnervation (TMR) cases for relief of neuroma and phantom limb pain: UK perspective. J Plast Reconstr Aesthet Surg. 2022 Mar;75(3):960-969. doi: 10.1016/j.bjps.2021.09.068. Epub 2021 Oct 22. PMID 34840118
- [Background] Cascini S, Agabiti N, Davoli M, Uccioli L, Meloni M, Giurato L, Marino C, Bargagli AM. Survival and factors predicting mortality after major and minor lower-extremity amputations among patients with diabetes: a population-based study using health information systems. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001355. doi: 10.1136/bmjdrc-2020-001355. PMID 32690575
- [Background] Gallizzi M, Gagnon C, Harden RN, Stanos S, Khan A. Medication Quantification Scale Version III: internal validation of detriment weights using a chronic pain population. Pain Pract. 2008 Jan-Feb;8(1):1-4. doi: 10.1111/j.1533-2500.2007.00163.x. PMID 18211588
- [Background] de Bruijn ME, Arts CH, van de Meent H, Frolke JP. Management of the sciatic nerve during transfemoral amputation: a survey of Dutch surgeons. J Cardiovasc Surg (Torino). 2020 Aug;61(4):467-470. doi: 10.23736/S0021-9509.19.10733-1. Epub 2019 Mar 27. PMID 30917649
- [Derived] Tendijck GAH, van Schaik J, Dijkman RR, Niesters M, van Zwet EW, van den Hout WB, Ploeg AJ, van Rijt WG, de Ruiter GCW, Coert JH, Duraku LS, Zuidam JM, van de Water W, Pondaag W, van der Krogt H, Groen JL; PreventPAP consortium. Prevention of postamputation pain with targeted muscle reinnervation (PreventPAP trial): protocol for a national, multicentre, randomised, sham-controlled trial. BMJ Open. 2025 Nov 4;15(11):e105053. doi: 10.1136/bmjopen-2025-105053. PMID 41248411
- See also: Study coordinating center — https://leidennervecenter.org/